CLINICAL TRIAL: NCT00530686
Title: Pancreatic Islet Cell Transplantation - A Novel Approach to Improve Islet Quality and Engraftment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: Baylor Health Care System (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 008-095
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Islet Cell Transplantation; Type 1 Diabetes
Keywords: Diabetes Mellitus; Hypoglycemia; Hyperglycemia; Type 1 Diabetes; Islet cell transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Hypoglycemia; Hyperglycemia | interventions — Islets of Langerhans Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Islet cell transplantation — The process is based on the enzymatic isolation of the pancreatic islets of Langerhans from an organ procured from a cadaveric donor; the islets obtained are injected into the liver of the recipient via percutaneous catheterization of the portal venous system . This procedure allows the selective transplantation of the insulin-producing cell population avoiding open surgery as well as the transplantation of the duodenum and the exocrine pancreas and their related morbidity.

SUMMARY:
The purpose of this study is to assess a novel approach to immunosuppression in allogenic pancreatic islet cell transplant recipients. In addition, the study aims to assess remote site islet processing with culture for pancreatic islet cell transplantation in human subjects.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) type I is a disease that has significant social and economical impact. The prevalence of the disease in the United States is about 120,000 in individuals aged 19 or less and 300,000 to 500,000 at all ages and 150 million worldwide.

So far there are no mechanical devices able to effectively adjust the dose of insulin injected according to the serum glucose in patients with DM. This leads to less than perfect sugar control, with episodes of hypoglycemia. Successful pancreas transplantation averts the need of insulin administration.

The emerging alternative to whole organ pancreas transplantation is pancreatic islet cell transplantation (ICT). The process is based on the enzymatic isolation of the pancreatic islets from an organ procured from a cadaver donor. The islets obtained are injected into the liver in the recipient via percutaneous catheterization of the portal venous system. This procedure allows the selective transplantation of the insulin-producing cell population avoiding open surgery as well as the transplantation of the duodenum and the exocrine pancreas and their related morbidity.

The initial efforts with ICT had only modest results. The immunosuppression regimen was similar to the one used in solid organ transplantation, based on high dose steroids and calcineurin inhibitors - both agents with diabetogenic effects. The results improved markedly with the changes in the manipulations of the islets, and the change in immunosuppression thus avoiding the higher doses of steroids and using sirolimus, tacrolimus and daclizumab initiated by the investigators group at the University of Alberta in Edmonton, Canada. Their protocol requires in general two islet cell infusions in order to attain the critical cell mass necessary to achieve insulin-independency. The changes in treatment were adopted as the Edmonton Protocol, which is used in several transplant centers, worldwide.

Isolation of the islets from donor pancreata will occur in the Baylor University Medical Center Islet Cell Processing Laboratory (ICPL). The islet cell infusion is performed in the Interventional Radiology Suite at Baylor University Medical Center or Baylor All Saints Medical Center by an interventional radiologist. The procedure takes place in a suite designed for invasive procedures using sterile technique with access to general anesthesia if necessary. Following the procedure the patient is observed in the Interventional Radiology recovery area for as long as necessary as determined by a Physician and then transferred to the Transplant Service for an overnight stay. After recovery, the patient is admitted to the hospital on the Transplant Service for a 1-2 day observation.

The focus of the research in the ICT is centered on the development of a safe and effective procedure that will eventually replace surgical pancreas transplantation together with an ideal immunosuppressive regimen that provides safe and effective prevention against rejection, while minimizing the adverse events associated that negatively impact transplant recipient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been fully informed and has signed an IRB approved informed consent form and is willing and able to follow study procedures for the full 24 months
* Patient is expected to receive an islet cell transplant (up to 3 infusions) for type I diabetes mellitus
* Type I diabetes mellitus of more than 5 years duration
* Age between 18 and 65
* Unstable diabetes mellitus control, as defined by glucose measurements above 200 mg/dL and/or below 80 mg/dL despite adequate medical care from a diabetology care team
* Hypoglycemia unawareness, as defined by episodes of loss of cognitive function; or the inability to recognize glucose levels below 50 mg/dL; or frequent episodes of symptomatic hypoglycemia; or admission to the hospital for hypo/hyperglycemic
* Incapacitating signs and symptoms, as defined by the referring physician
* HbA1c > 6.5
* Psychogenically able to comply, in the opinion of the investigator
* Female patients of childbearing potential must have a negative urine or serum pregnancy test upon hospitalization or within 7 days prior to enrollment and have agreed to utilize effective birth control throughout the study as well as for 6 weeks following study completion.

Exclusion Criteria:

* Patient has previously received or is receiving an organ or bone marrow transplant
* Patient has a known hypersensitivity to Tacrolimus, sirolimus, dacluzimab, or CellCept
* Patient is pregnant or lactating
* Patient has participated in a blinded trial or participated in a trial involving a non-marketed (investigational) drug within 3 months of enrollment
* Patient has participated in a trial involving a marketed drug or an infusion device within 30 days of the start of the trial
* Glofil or Creatinine Clearance < 60 mL/min
* Serum Creatinine > 1.6 mg/dL consistently
* Body mass index > 28
* Malignancy other than basal cell carcinoma or squamous cell carcinoma
* Radiographic evidence of pulmonary infection
* Evidence of liver disease as evidenced by >2X ULN for AST, ALT, Alk Phos., or T bili.
* Active infections
* Hypercoagulable states (history of recurrent venous thrombosis, defined thrombophilia)
* Bleeding / coagulation disorders
* Basal C-Peptide > 0.3 ng/dL
* HbA1c > 12%
* Insulin requirement >0.7 IU/kg/day
* Seropositivity for HIV, HBV, HCV, HTLV-1
* Abnormal Pap smear, active gynecological infection
* Positive exercise or chemical tolerance test
* Patients currently under treatment for a medical condition requiring chronic use of steroids at a dose of prednisone >5mg/day will be excluded
* Substance/alcohol abuse
* Untreated proliferating diabetic retinopathy
* PPD conversion or positive PPD without INH
* No Primary care physician or primary care physician less than 6 months
* Smoking in the last 6 months
* Abnormal CBC / Hemoglobin < 12 g/dL
* Macroalbuminuria > 300 mg/24 hours
* Untreated hyperlipidemia - TC > 200 mg/dL, TGC > 200 mg/dL, LDL > 130 mg/dL
* Untreated hyponatremia, hypokalemia, hypercalcemia, hypocalcemia
* Iodine contrast allergy
* PSA > 4
* PRA > 20%
* Active peptic ulcer disease/gallstones/hemangioma
* Abnormal mammogram

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
1)Presence or absence of hypoglycemic unawareness 2) To assess incidence of hypoglycemic episodes 3) To assess insulin requirements in patients who did not become insulin independent. | 24 months

SECONDARY OUTCOMES:
To assess the achievement of insulin independence at 12 month and 24 month post transplant in patients who underwent allo islet cell transplantation. | 12 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Onaca, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Annette C. & Harold C. Simmons Transplant Institute - Baylor University Medical Center, Dallas Texas, USA - Baylor All Saints Medical Center, Fort Worth Texas, USA, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided